CLINICAL TRIAL: NCT00782015
Title: Effects of Almonds on Vascular Reactivity and Biomarkers of Inflammation, Oxidative Stress and Endothelial Function in Patients With Coronary Artery Disease
Brief Title: Effects of Almonds on Vascular Reactivity in Patients With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Jeffrey Blumberg, PI, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TuftsIRB8723
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Vascular Disease; Endothelial Dysfunction; Heart Disease; Cardiovascular Diseases; Hypertension
Keywords: almonds; heart disease; vascular reactivity; inflammation; dyslipidemia; oxidative stress
MeSH Terms: conditions — Vascular Diseases; Heart Diseases; Cardiovascular Diseases; Hypertension; Inflammation; Dyslipidemias | interventions — Nuts

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- almonds (Active Comparator): 3 oz/d almonds
  Interventions: Dietary Supplement: Almonds
- Placebo (Placebo Comparator): NCEP Step 2 diet
  Interventions: Dietary Supplement: Placebo Comparator:

INTERVENTIONS:
Dietary Supplement: Almonds — 3 oz. of almonds per day, supplied as 1 oz. snack packs to be consumed for 6 weeks.
  Other Names: Nuts
  Arms: almonds
Dietary Supplement: Placebo Comparator: — NCEP Step 2 diet
  Arms: Placebo

SUMMARY:
This is a study of the effects of 3 oz almonds added daily to a National Cholesterol Education Program Therapeutic Lifestyle Changes (TLC) diet in improving endothelial function in patients with Coronary Artery Disease. The study seeks to determine if these effects are mediated via an increase in Nitric Oxide synthesis and reductions in dyslipidemia and systemic inflammation.

Vascular reactivity will be assessed via flow mediated dilation with endothelium-independent and hyperemic flow measured in the right brachial artery by non-invasive 2-dimensional and Doppler ultrasound. Serum will be collected and analyzed for biomarkers of dyslipidemia, inflammation, endothelial function, vascular reactivity and oxidative stress.

DETAILED DESCRIPTION:
The study is a randomized, crossover, 6 week intervention trial design with a 6 week run in on the TLC diet and a 6 week washout on the TLC diet between control and intervention periods. Forty subjects with verified and stable coronary artery disease will be enrolled in the study. The control intervention involved maintaining a steady TLC diet without nuts which will be monitored with counseling and dietary assessments. The almond intervention involved consuming 3 oz. of almonds per day and adjusting lipid intake to remain isocaloric with the TLC diet alone. Again subjects will be monitored with counseling and dietary assessments.

At the beginning and end of each intervention period subjects will be tested for endothelial function using flow mediated dilation and blood and urine samples will be collected for biochemical analysis for markers of inflammation, dyslipidemia, and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Stable CAD Patients (men & postmenopausal women)
* aged 20-80 years
* weighing less than 115 Kg (BMI range 18.5-35 kg/m2)
* with coronary artery disease defined by the presence of lesions on coronary angiography, history of myocardial infarction, or positive stress test.
* Subjects are eligible to participate after a stent procedure only after they have been stable for one month after the stent procedure.
* All Ethnic Groups.
* Languages: English

Exclusion Criteria:

* Subjects with heart failure are not eligible for participation in this study.
* History or known allergy to nuts of any kind
* Women with a positive urine beta HCG pregnancy test and lactating women or women who are planning to become pregnant.
* Regular consumption of ≥ 5 oz nuts/week for 6 weeks prior to study admission
* Clinical history of other major illness including end-stage cancer, renal failure, hepatic failure, gastrointestinal disorders that may impair absorption, or other conditions that in the opinion of the principal investigator make a clinical study inappropriate.
* Regular use of oral steroids
* Cigarette smoking and/or nicotine replacement use
* Regular daily intake of ≥ 2 alcoholic drinks
* Illicit drug use
* History of a psychological illness or condition such as to interfere with the subject's ability to understand the requirements of the study.
* No dietary supplements containing phenolic compounds, i.e., herbal preparations, or berry containing preparations (such as cranberry capsules) for one month prior to study admission.
* Treatment with an investigational new drug within the last 30 days.
* Treatment with Vitamin E, Vitamin C, beta carotene, lipoic acid, or other food or herbal supplements within 1 month of enrollment (subjects taking multivitamins or other forms of vitamin E and C in doses that do not exceed two times the RDA will not be excluded).
* The following medications will be withheld in the morning of each ultrasound study visit as follows:

All vasoactive medications (nitrates, calcium channel blockers, beta blockers, angiotensin converting enzyme inhibitors, and other vasodilators). Subjects will take their medications immediately after the ultrasound measurements are taken.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Endothelial Function as determined by flow mediated dilation and and biochemical markers of endothelial function. | After 6 weeks eating almonds

SECONDARY OUTCOMES:
Biochemical markers of inflammation, such as cytokines | After 6 weeks of eating almonds
Biochemical markers of dyslipidemia, such as lipid profiles | After 6 weeks of eating almonds
Biomarkers of oxidative stress, such as isoprostanes and 8OHdG | After 6 weeks of eating almonds

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Blumberg, PhD, Principal Investigator — HNRCA Tufts University; Joseph Vita, MD, Principal Investigator — Boston University
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University (HNRCA), Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chen CY, Holbrook M, Duess MA, Dohadwala MM, Hamburg NM, Asztalos BF, Milbury PE, Blumberg JB, Vita JA. Effect of almond consumption on vascular function in patients with coronary artery disease: a randomized, controlled, cross-over trial. Nutr J. 2015 Jun 17;14:61. doi: 10.1186/s12937-015-0049-5. PMID 26080804